CLINICAL TRIAL: NCT01141348
Title: Intensive Behavioral Weight Management in Public Health Settings: Weight-Wise
Brief Title: The Weight-Wise Weight Loss Translation Study
Acronym: Weight-Wise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Davidson County Health Department (Unknown); Forsyth County Health Department (Unknown); Lincoln County Health Department (Unknown); Nash County Health Department (Unknown); Albemarle Regional Health Services (Unknown); Warren County Health Department (Unknown)
Responsible Party: Carmen Samuel-Hodge, PhD, MS, RD, University of North Carolina - Center for Health Promotion and Disease Prevention
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08-0055
Record Dates: First submitted 2010-05-06; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Overweight; Obesity; Cardiovascular Disease
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Special Intervention (Experimental)
  Interventions: Behavioral: Special Intervention
- Delayed Intervention (Experimental)
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: Special Intervention — 16 week behavioral weight loss intervention included 2 hour weekly group sessions
  Arms: Special Intervention
Behavioral: Delayed Intervention — During the randomized controlled trial, the Delayed Intervention (DI) group received two newsletters with study updates and general health information. Following the trial, the DI group received a 10-week weight loss program.
  Arms: Delayed Intervention

SUMMARY:
The overall goal of the translational research is to evaluate the processes and outcomes of implementing, in a range of public health agencies, an intense, evidence-based behavioral weight loss intervention with demonstrated effectiveness among midlife low-income women. The intervention was originally studied in a single coordinated community health care center/church setting and delivered by research staff. The investigators will evaluate the intervention's translation and test its effectiveness as implemented by existing staff in six public health agencies supported by local community resources.

DETAILED DESCRIPTION:
Low-income women in the US have the highest rates of overweight and obesity, putting them at increased risk for diabetes, heart disease, and other chronic illnesses. Because mean body mass index gradually increases during adult life and peaks at 50-59 years of age, low income women between 40-64 years are a group deserving of special attention. While there is sufficient evidence that some behavioral weight management interventions are effective in producing clinically meaningful levels of weight loss with reductions in cardiovascular risk factors and delayed onset of diabetes, there is a research gap in translating these efficacious interventions to real life settings and diverse population groups. Research that seeks to translate effective behavioral weight management interventions from resource-intensive efficacy trials to long-term adoption and implementation by public health settings serving a diverse low-income population is timely and of great public health significance. This translational research can provide important information to decision-makers about evidence-based intervention delivery, resource allocation, and workforce preparation.

The overall goal of the proposed research is to evaluate the processes and outcomes of translating from research to practice an intense, evidence-based behavioral weight loss intervention with demonstrated effectiveness among midlife low-income women. Originally studied in a single coordinated community health care center/church setting and delivered by research staff (Weight-Wise Pilot Study), we will evaluate the translation of and test the effectiveness of this intervention as implemented by existing staff in a range of county health departments supported by local community resources.

To evaluate the translation process, we will use the RE-AIM framework, diffusion of innovation theory, and systematic models of adaptation to assess: 1) factors related to reach; contextual or setting-specific factors necessary for successful adoption and implementation; 2) effectiveness of facilitator training and stakeholder collaborations; 3) adaptation and fidelity during implementation; and 4) costs associated with the implementation and outcomes. To test the intervention's effectiveness, we will enroll 240 overweight or obese low-income women, 40-64 years of age, at 6 representative public health agencies. Participants will be randomized to receive a 16-week behavioral weight loss intervention (special intervention group) or usual care (wait listed control group). The primary study outcome at 5 month follow-up is weight change; secondary outcomes include change in blood pressure, dietary intake, physical activity, and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between 27.5 and 45
2. willing to lose 5% or more of initial body weight and follow recommendations for healthy dietary and PA patterns
3. English-speaking
4. able and willing to give informed consent
5. household income less than or equal to 250% of federal poverty guidelines.

Exclusion Criteria:

1. medical or physical limitations to engaging in moderate level physical activity
2. medical or other contraindications to weight loss
3. history of gastric bypass surgery or scheduled surgery for this purpose
4. weight loss of > 20 lbs in the last 3 months
5. current use of medication for weight loss
6. treatment of psychosis
7. diagnosis of Type 1 diabetes.

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Weight Change difference between baseline and 4 month follow-up | Baseline and 4 month follow-up

SECONDARY OUTCOMES:
Change in blood pressure, dietary intake, physical activity, and quality of life between baseline and 4 month follow-up | Baseline and 4 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Samuel-Hodge, PhD, MS, RD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (6):
- United States (6):
  - Albemarle Regional Health Services, Elizabeth City, North Carolina
  - Davidson County Health Department, Lexington, North Carolina
  - Lincoln County Health Department, Lincolnton, North Carolina
  - Nash County Health Department, Nashville, North Carolina
  - Warren County Health Department, Warrenton, North Carolina
  - Forsyth County Health Department, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Jones SA, Evenson KR, Johnston LF, Trost SG, Samuel-Hodge C, Jewell DA, Kraschnewski JL, Keyserling TC. Psychometric properties of the modified RESIDE physical activity questionnaire among low-income overweight women. J Sci Med Sport. 2015 Jan;18(1):37-42. doi: 10.1016/j.jsams.2013.12.007. Epub 2014 Jan 1. PMID 24462117